CLINICAL TRIAL: NCT00232297
Title: Double Blind Placebo Controlled Dose Ranging Study of the Efficacy and Safety of SSR149744C 100 OR 300 mg for the Prevention of Ventricular Arrhythmia-Triggered ICD Interventions
Acronym: ICARIOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5349
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Arrhythmia; Tachycardia, Ventricular; Ventricular Fibrillation
Keywords: Tachycardia, Ventricular; Ventricular Fibrillation; Defibrillators Implantable; Arrhythmia; Anti-arrhythmia agents
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — celivarone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SSR149744C

SUMMARY:
Primary objective:

* to assess the efficacy of SSR149744C for the prevention of ventricular arrhythmia-triggered ICD interventions.

Secondary objectives:

* to assess versus placebo the tolerability of the different dose regimens of SSR149744C in the selected population.
* to document SSR149744C plasma level during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an ICD implanted during the previous year for documented spontaneous life-threatening ventricular arrhythmia OR implanted with an ICD and with at least one appropriate ICD therapy (shock or anti-tachycardia pacing) for ventricular tachycardia or ventricular fibrillation in the previous year.
* Left ventricular ejection fraction measured by 2D-echocardiography must have been documented to be less than 40% in the last 6 months.

Exclusion Criteria:

MAIN CRITERIA (non-exhaustive list):

* Women of childbearing potential without adequate birthcontrol, Pregnant Women, Breastfeeding women, conditions which increase the risk of severe antiarrhythmic drug side effects, severe associated conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2005-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is time to all ventricular tachycardia or ventricular fibrillation arrhythmia leading to any ICD intervention (anti-tachycardia pacing or ICD shock).

SECONDARY OUTCOMES:
Time to all arrhythmia episodes leading to at least one documented ICD shock.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Result] Gojkovic O, Aliot EM, Capucci A, Connolly SJ, Crijns H, Hohnloser SH, Kulakowski P, Roy D, Radzik D, Singh BN, Kowey PR. Celivarone in patients with an implantable cardioverter-defibrillator: adjunctive therapy for the reduction of ventricular arrhythmia-triggered implantable cardioverter-defibrillator interventions. Heart Rhythm. 2012 Feb;9(2):217-224.e2. doi: 10.1016/j.hrthm.2011.09.073. Epub 2011 Oct 4. PMID 21978965
- See also: Related Info — http://www.sanofi-aventis.com